CLINICAL TRIAL: NCT06947629
Title: Role of Frozen Section in Categorization of Thyroid Follicular Neoplasm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Sayed, Demonstrator at Pathology Department In New Valley University, New Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-2025-201196
Record Dates: First submitted 2025-04-07; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Role of Frozen Section in Categorization of Thyroid Follicular Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Evaluation Group (Experimental)
  Interventions: Diagnostic Test: Intraoperative Frozen Section

INTERVENTIONS:
Diagnostic Test: Intraoperative Frozen Section — Intraoperative Frozen Section analysis which will include the following steps:
  - The specimen will undergo both gross and microscopic examination:
  1. Gross examination: Evaluation of nodular features including, multiplicity, size, outlines, color and consistency.
  2. Microscopic examination: Assessment of capsular pattern, capsular invasion, thickness of capsule, vascular invasion and number of invaded vessels and the presence or absence of papillary structures.

SUMMARY:
The goal of this prospective study is to assess the effectiveness of frozen section in distinguishing between benign and malignant tumors in the category of follicular thyroid neoplasm to prevent over-surgery for benign follicular neoplasm (lobectomy Vs total thyroidectomy).

The main questions, it aims to answer are:

The follicular neoplasm is benign or malignent? how far is FNAC valid and accurate? Researchers will compare the results of frozen section and paraffin embedded sections to evaluate the validity and accuracy of FNAC.

DETAILED DESCRIPTION:
Thyroid tumors are the most common endocrine neoplasms, with their incidence steadily rising over the past few decades, reaching approximately 8.7 cases per 100,000 people annually in Europe. The majority of thyroid tumors are benign accounting for over 90% of cases, whereas malignant thyroid tumors are relatively less common. Thyroid cancer represents 1-2% of all newly diagnosed malignancies worldwide, with papillary thyroid carcinoma (PTC) being the most prevalent (80%) followed by follicular thyroid carcinomas (FTC) (15%). Fine needle aspiration cytology (FNAC) is the primarily diagnostic tool for thyroid nodule. However, its accuracy in distinguishing between benign and malignant follicular neoplasms is limited, necessitating further histopathological evaluation. The Bethesda system classifies FNAC results into six categories, with follicular neoplasm/suspicious for follicular neoplasm (category IV) carrying a moderate risk of malignancy. Differentiating between benign and malignant follicular neoplasms requires assessing capsular and vascular invasion. Intraoperative frozen section (FS) has been used for decades to provide rapid histologic assessment guiding the extent of surgery (lobectomy Vs total thyroidectomy). However, its utility remains controversial due to variability in diagnostic accuracy and cost-effectiveness. The recent 5th edition of the WHO classification (2023) categorizes follicular-derived thyroid tumors into benign, low-risk and malignant neoplasms, further refining diagnostic criteria. This study aims to evaluate the accuracy of FNAC and FS in diagnosing follicular thyroid neoplasms, optimizing surgical decisions and reducing unnecessary total thyroidectomies in benign cases.

ELIGIBILITY:
Inclusion Criteria:

* Cases presented with a thyroid nodule, diagnosed as "follicular neoplasm" (Bethesda category IV) by fine needle aspiration cytology, and underwent hemi-thyroidectomy.

Exclusion Criteria:

* Cases with thyroid nodule and diagnosed by fine needle aspiration cytology as non-neoplastic lesions, suspicious for malignancy or as malignant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Role of frozen section evaluation in the diagnosis of malignant follicular neoplasm from benign in Thyroid Follicular Neoplasm | two weeks
  Role of frozen section evaluation in the diagnosis of malignant follicular neoplasm from benign.

SECONDARY OUTCOMES:
Assessment of the accuracy of fine needle aspiration cytology in diagnosis of follicular neoplasm. | three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Howayda I Hassan, professor, Study Chair — Faculty of Medicine, Assiut Universiy, Assiut, Egypt; Mahmoud F Sherif, Assistant Professor, Study Director — Faculty of Medicine, Assiut Universiy, Assiut, Egypt
Locations (1):
- Assiut Universiy Hospital and Private pathology laboratory, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Data is available with the corresponding offer on reasonable request